CLINICAL TRIAL: NCT03659214
Title: Impact of the Introduction of ORKAMBI on Anxiety, Depression, Quality of Life and Adherence of Adolescents and Young Adults
Acronym: ORK-AJA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: VERTEX Pharmaceutical (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180003; 2018-A01561-54 (Other: ID-RCB)
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Orkambi; Adherence; Adolescent; Anxiety; Depression; Psychology
MeSH Terms: conditions — Cystic Fibrosis; Anxiety Disorders; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated group: Patients with proven CF (sweat-test > 60 mEq, 2 DF508 CF causing mutations, 12 to 20 years, and treated with ORKAMBI)
  Interventions: Behavioral: Questionnaires
- Control group: Patients not carrying 2 DF508 CF causing mutations, not treated with ORKAMBI, and not carrying the G551D, G178R, S549N, S549R, G551S, G1244E,S1251N, S1255P or G1349D mutation or treated with Kalydeco
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Answering 4 questionnaires : anxiety, depression, quality of life and adherence

SUMMARY:
The aim of this project is to evaluate the psychological reshuffle induced by ORKAMBI. The particular focus of this study is the consequence of its introduction on anxiety, depression, quality of life and adherence to all cystic fibrosis (CF) treatment. To answer this question investigators will monitor the psychological function of CF adolescents and young adults treated with ORKAMBI and compare them to CF adolescents and young adults not treated with ORKAMBI.

DETAILED DESCRIPTION:
Introduction of KALYDECO then ORKAMBI, as a personalized medicine in the therapeutic strategy of Cystic Fibrosis (CF) may deeply modify the prognosis of patients with CF. These approaches realize the dream of short-circuiting the molecular mechanism of the disease and therefore opens the perspective of an extended and functional survival. It suddenly offers the possibility of a completely new future to the patient and his family, and therefore must deeply impact on the psychological function of all involved. Moreover, those new therapies may also modify the adherence to CF basic treatment, as it brings a new feeling of good health and the hope of a longer life. For that reason there is a need to investigate modifications of the psychological state of mind induced by the treatment with ORKAMBI in CF adolescents and young adults.

This project aims to understand the psychological impact and to study the consequences of the introduction of ORKAMBI on adherence to CF treatment, anxiety, depression and quality of life.

To answer this question, investigators will evaluate the psychological function of adolescents and young adults, aged 12 to 20 years, with CF treated with ORKAMBI, and compare it to other adolescents and young CF adults not treated with ORKAMBI.

This is a cohort prospective study, with a 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Treated group: Patients with proven CF (sweat-test > 60 mEq, 2 DF508 CF causing mutations, 12 to 20 years, and treated with ORKAMBI
* Control group: Patients not carrying 2 DF508 CF causing mutations, not treated with ORKAMBI, and not carrying the G551D, G178R, S549N, S549R, G551S, G1244E,S1251N, S1255P or G1349D mutation or treated with Kalydeco

Exclusion Criteria:

* Transplanted patients
* Patients younger than 12 years
* Patients older than 20 years

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: CF Center patients
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Score of Generalized Anxiety Disorder-7 questionnaire (GAD-7) | 24 months
  to assess the impact on Anxiety

SECONDARY OUTCOMES:
Score of Patient Health Questionnaire-9 (PHQ-9 ) | 24 months
  To assess the impact on Depression
Scores of Cystic Fibrosis Questionnaire 14+ (CFQ 14+) | 24 months
  Disease-specific instrument designed to measure impact on overall health, daily life, perceived well-being and symptoms (Quality of Life)
GIRERD Scale | 24 months
  The 6 items are assessed using a YES/NO answer .The scale was validated in patients with chronic disease to assess medication adherence

CONTACTS AND LOCATIONS:
Overall Officials: Maya KIRSZENBAUM, Psychologist, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Pneumology -CRCM - Necker - Enfants maladies Hospital (AP-HP), Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pendleton DA, David TJ. The compliance conundrum in cystic fibrosis. J R Soc Med. 2000;93 Suppl 38(Suppl 38):9-13. No abstract available. PMID 10911813
- [Background] Bucks RS, Hawkins K, Skinner TC, Horn S, Seddon P, Horne R. Adherence to treatment in adolescents with cystic fibrosis: the role of illness perceptions and treatment beliefs. J Pediatr Psychol. 2009 Sep;34(8):893-902. doi: 10.1093/jpepsy/jsn135. Epub 2009 Feb 5. PMID 19196850
- [Background] Zindani GN, Streetman DD, Streetman DS, Nasr SZ. Adherence to treatment in children and adolescent patients with cystic fibrosis. J Adolesc Health. 2006 Jan;38(1):13-7. doi: 10.1016/j.jadohealth.2004.09.013. PMID 16387243
- [Background] Butner J, Berg CA, Osborn P, Butler JM, Godri C, Fortenberry KT, Barach I, Le H, Wiebe DJ. Parent-adolescent discrepancies in adolescents' competence and the balance of adolescent autonomy and adolescent and parent well-being in the context of Type 1 diabetes. Dev Psychol. 2009 May;45(3):835-49. doi: 10.1037/a0015363. PMID 19413435
- [Background] Arias Llorente RP, Bousono Garcia C, Diaz Martin JJ. Treatment compliance in children and adults with cystic fibrosis. J Cyst Fibros. 2008 Sep;7(5):359-67. doi: 10.1016/j.jcf.2008.01.003. Epub 2008 Mar 4. PMID 18304896
- [Background] Marciel KK, Saiman L, Quittell LM, Dawkins K, Quittner AL. Cell phone intervention to improve adherence: cystic fibrosis care team, patient, and parent perspectives. Pediatr Pulmonol. 2010 Feb;45(2):157-64. doi: 10.1002/ppul.21164. PMID 20054860
- [Background] Blackwell LS, Marciel KK, Quittner AL. Utilization of patient-reported outcomes as a step towards collaborative medicine. Paediatr Respir Rev. 2013 Sep;14(3):146-51. doi: 10.1016/j.prrv.2013.04.003. Epub 2013 May 27. PMID 23721854
- [Background] Girerd X, Radauceanu A, Achard JM, Fourcade J, Tournier B, Brillet G, Silhol F, Hanon O. [Evaluation of patient compliance among hypertensive patients treated by specialists]. Arch Mal Coeur Vaiss. 2001 Aug;94(8):839-42. French. PMID 11575214
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941